CLINICAL TRIAL: NCT07209618
Title: Rehabilitation of Alveolar Horizontal Bone Deficiencies Using Autogenous Onlay Bone Grafting With Simultaneous Implant Placement: A Novel Approach
Brief Title: Horizontal Ridge Augmentation With Simultaneous Implant Placement Using Autogenous Ramus Grafts
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Oznur Ozalp, Principal Investigator, Akdeniz University
Other Study IDs: AKDENIZ-RAMUS-2018-TBAEK-415
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Bone Loss; Tooth Loss / Rehabilitation
MeSH Terms: conditions — Alveolar Bone Loss; Tooth Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Simultaneous implant + ramus graft group
  Interventions: Procedure: utogenous mandibular ramus block grafting with simultaneous dental implant placement; Procedure: Autogenous mandibular ramus block graft with simultaneous implant placement

INTERVENTIONS:
Procedure: utogenous mandibular ramus block grafting with simultaneous dental implant placement — Horizontal alveolar ridge augmentation performed using autogenous block grafts harvested from the mandibular ramus. The graft was fixed to reconstruct the buccal wall, followed by immediate placement of dental implants in the same surgical session. Prosthetic loading was initiated 4 months postoperatively.
Procedure: Autogenous mandibular ramus block graft with simultaneous implant placement — Horizontal alveolar ridge augmentation performed using autogenous block grafts harvested from the mandibular ramus. The graft was fixed to reconstruct the buccal wall, followed by immediate placement of dental implants in the same surgical session. Prosthetic loading was initiated 4 months postoperatively.

SUMMARY:
This retrospective observational study evaluated the clinical outcomes of simultaneous implant placement with horizontal ridge augmentation using autogenous mandibular ramus block grafts. Sixteen patients were treated between January 2018 and March 2025. Clinical and radiological data were analyzed to assess implant survival, osseointegration, and graft incorporation.

DETAILED DESCRIPTION:
Horizontal alveolar bone deficiency is a significant challenge in implant rehabilitation. Traditional staged augmentation techniques prolong treatment time and increase morbidity. This study introduces a novel approach in which autogenous mandibular ramus block grafts were used to reconstruct buccal walls simultaneously with implant placement. Sixteen patients received 23 implants. Outcomes included implant survival, osseointegration success, bone healing, and complications during a mean follow-up of 30.6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* ASA I or II status
* Presence of horizontal alveolar ridge deficiency requiring augmentation for implant placement
* Treated with autogenous mandibular ramus block grafts and simultaneous implant placement
* Provided informed consent for surgical and prosthetic procedures, and use of clinical and radiological data

Exclusion Criteria:

* Systemic conditions interfering with dental implant treatment (e.g., uncontrolled diabetes, metabolic bone disease)
* Incomplete clinical or radiological records
* Patients with contraindications for oral surgical procedures
* Patients unwilling to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sixteen patients (9 females, 7 males; mean age 41.4 years, range 21-61 years) with horizontal alveolar ridge deficiencies were treated at the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Akdeniz University, between January 2018 and March 2025. All patients underwent horizontal ridge augmentation with autogenous mandibular ramus block grafts in conjunction with simultaneous implant placement.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
implant survival rate | 4 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ozalp, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided